CLINICAL TRIAL: NCT02805504
Title: Efficacy of the Liposomal Bupivacaine for Postoperative Pain Control in Urologic Procedures
Brief Title: Liposomal Bupivacaine for Postoperative Pain Control in Urologic Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, D. Duane Baldwin, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5160165
Record Dates: First submitted 2016-06-14; First posted 2016-06-20 (Estimated); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Diseases
Keywords: Bupivacaine; Minimally Invasive Surgical Procedures
MeSH Terms: conditions — Urologic Diseases | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Experimental): This arm will receive intraoperative local Liposomal Bupivacaine injection (Exparel) at the port placement site.
  Interventions: Drug: Exparel
- Marcaine (Active Comparator): This group will receive will local bupivacaine HCl (Marcaine) injection at the port placement site.
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Exparel — This group will receive intraoperative local Liposomal Bupivacaine injection at the surgical site.
  Other Names: liposomal bupivacaine
  Arms: Exparel
Drug: Marcaine — This group will receive intraoperative Bupivacaine HCl injection at the surgical site.
  Other Names: Bupivacaine HCl
  Arms: Marcaine

SUMMARY:
A prospective, randomized controlled study to determine the efficacy of liposomal bupivacaine given by local injection at all the wound sites in patients undergoing urologic surgeries.

DETAILED DESCRIPTION:
A prospective, randomized controlled study to determine the efficacy of liposomal bupivacaine given by local injection at all the wound sites in patients undergoing urologic surgeries. Subjects of prospective study will be randomly divided using electronic program into two groups:

The first group will receive intraoperative local Liposomal Bupivacaine injection at the port placement site. The control group will receive will local Marcaine (bupivacaine HCl) injection

Primary Outcome Measures:

* Total opioid consumption measured in intravenous morphine equivalents dose during the postoperative hospital Stay
* Postoperative pain assessment using visual Analog Pain Scores & Brief Pain Inventory form.
* Length of Hospital Stay
* Time to First Opioid Use.
* Postoperative Constipation , paralytic ileus

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urologic surgery.

Exclusion Criteria:

* Pregnant and/or nursing mothers.
* Allergy to bupivacaine.
* History of drug/alcohol abuse.
* Severe cardiovascular, hepatic, renal disease or neurological impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Keheila, MD, Study Director — Loma Linda University Medical Center
Locations (1):
- Loma Linda Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelsattar JM, Boughey JC, Fahy AS, Jakub JW, Farley DR, Hieken TJ, Degnim AC, Goede W, Mohan AT, Harmsen WS, Niesen AD, Tran NV, Bakri K, Jacobson SR, Lemaine V, Saint-Cyr M. Comparative Study of Liposomal Bupivacaine Versus Paravertebral Block for Pain Control Following Mastectomy with Immediate Tissue Expander Reconstruction. Ann Surg Oncol. 2016 Feb;23(2):465-70. doi: 10.1245/s10434-015-4833-4. Epub 2015 Aug 26. PMID 26307232
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] White S, Vaughan C, Raiff D, Eward W, Bolognesi M. Impact of liposomal bupivacaine administration on postoperative pain in patients undergoing total knee replacement. Pharmacotherapy. 2015 May;35(5):477-81. doi: 10.1002/phar.1587. Epub 2015 May 4. PMID 25940854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel | Marcaine
Started | 63 | 73
Completed | 63 | 73
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Marcaine | Total
Number analyzed (Participants) | 63 | 73 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 38 | 68
  >=65 years | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.3) | 62.7 (10.7) | 62.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 23 | 25 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 63 | 73 | 136
Region of Enrollment [Number; unit: participants]
  United States | 63 | 73 | 136

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption
Description: Postoperative analgesic use will be measured in oral morphine equivalents dose given to patients in the first three days postoperatively
Time Frame: Postoperative days 1-3
Population: During an audit by the compliance department of Loma Linda University, it was noted that some consents were incomplete and therefore could not undergo further analysis. Data presented has been taken from abstracts with preliminary analyses presented prior to the audit and subsequently should be interpreted with caution.
Measure: Mean (Standard Deviation); unit: morphine equivalent
Groups:
- Exparel: This arm will receive intraoperative local Liposomal Bupivacaine injection (Exparel) at the port placement site.
  Exparel: This group will receive intraoperative local Liposomal Bupivacaine injection at the surgical site.
  No reportable study outcome data is available per IRB determination after study closure.
- Marcaine: This group will receive will local bupivacaine HCl (Marcaine) injection at the port placement site.
  Marcaine: This group will receive intraoperative Bupivacaine HCl injection at the surgical site.
  No reportable study outcome data is available per IRB determination after study closure.
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 53 | 55
morphine equivalent | 16.4 (19.4) | 15.3 (16.2)

2. Primary Outcome: Postoperative Pain Assessment
Description: Pain score (0-10) will be used. This will be based on a standard visual analog scale, where 0 indicates no pain and 10 indicates the most severe pain reported by patients.
Time Frame: Postoperative day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 53 | 55
units on a scale | 4.6 (2.1) | 4.6 (2.4)

3. Primary Outcome: Length of Hospital Stay
Description: Duration of hospital stay after the surgery until time of discharge
Time Frame: Duration of stay in hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 53 | 55
Hours | 37 (31.8) | 36 (24)

4. Primary Outcome: Postoperative Complications
Description: Any complication related to the surgery within 30 days
Time Frame: 30 days postoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Marcaine
Number analyzed (Participants) | 53 | 55
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 30-days postoperatively
Arm/Group | Exparel | Marcaine
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/73
Serious Adverse Events (participants affected / at risk) | 6/63 | 6/73
Other Adverse Events (participants affected / at risk) | 0/63 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel (N=63) | Marcaine (N=73)
Postoperative Ileus (Gastrointestinal disorders) | 4 | 4 — Postoperative ileus managed conservatively
Postoperative Bleeding (Surgical and medical procedures) | 1 | 0 — Postoperative bleeding requiring blood transfusion
Postoperative Hypotension (Surgical and medical procedures) | 1 | 1 — Postoperative hypotension or dehydration requiring fluid management
Stricture (Renal and urinary disorders) | 0 | 1 — Postoperative stricture requiring dilation

LIMITATIONS AND CAVEATS:
During an audit by the compliance department of Loma Linda University, it was noted that some consents were incomplete and therefore could not undergo further analysis. Data presented has been taken from abstracts with preliminary analyses presented prior to the audit and subsequently should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02805504/Prot_SAP_000.pdf